CLINICAL TRIAL: NCT05399082
Title: A Study to Evaluate the Feasibility of Robotic Bronchoscopy-guided Miniature Cryoprobe Biopsy of Peripheral Pulmonary Lesions
Brief Title: Feasibility of Performing Peripheral Pulmonary Lesion Biopsy Using Robotic Bronchoscopy-Guided Cryoprobe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Erbe USA Incorporated (Other)
Responsible Party: Principal Investigator, Ryan M. Kern, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 21-008716
Record Dates: First submitted 2022-05-20; First posted 2022-06-01 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Bronchi--Diseases; Lung Diseases, Obstructive; Lesions Mass
MeSH Terms: conditions — Bronchial Diseases; Lung Diseases, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard forceps biopsy then research cryoprobe biopsy (Experimental): Subjects scheduled for a biopsy of lung lesions using robotic bronchoscopy as part of their standard of care will have the lung lesion biopsied using forceps first followed by cryoprobe.
  Interventions: Device: Cryoprobe biopsy; Procedure: Forceps biopsy
- Research cryoprobe biopsy then standard forceps biopsy (Experimental): Subjects scheduled for a biopsy of lung lesions using robotic bronchoscopy as part of their standard of care will have the lung lesion biopsied using the cryoprobe first followed by forceps.
  Interventions: Device: Cryoprobe biopsy; Procedure: Forceps biopsy

INTERVENTIONS:
Device: Cryoprobe biopsy — A 1.1mm disposable cryoprobe that is passed through the working channel of the Ion Robotic bronchoscope to collect biopsy tissue
Procedure: Forceps biopsy — Biopsy forceps used to collect tissue

SUMMARY:
This research is being done to evaluate the feasibility, and biopsy quality, of using a 1.1mm disposable cryoprobe that is passed through the working channel of the Ion Robotic bronchoscope to collect biopsy tissue.

ELIGIBILITY:
Inclusion Criteria:

- Patient clinically meets indication for peripheral lung nodule biopsy and has been scheduled for robotic bronchoscopy.

Lesion Criteria:

- Pulmonary nodules of 8-50mm in largest dimension.

Exclusion Criteria:

* Patients with known bleeding diathesis; Platelet count < 50,000.
* Current use of systemic anticoagulation or antiplatelet therapy without the ability to hold therapy for the recommended amount of time prior to an invasive procedure (aspirin monotherapy is acceptable).
* Inability or unwillingness to give informed consent.
* Pregnant or nursing females, or females of child-bearing potential who decline a pregnancy test prior to enrollment.
* Pulmonary hypertension, defined as a right ventricular systolic pressure > 50 mmHg.
* Individuals with current or recent systematic conditions, such as, acute kidney injury, or conditions that would mandate anticoagulation, such as a recent coronary stent.
* International Normalized Ratio (INR) < 1.5.
* Do Not Resuscitate (DNR) status; Do Not Intubate (DNI) status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2023-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Kern, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Forceps Biopsy First, Then Research Cryoprobe Biopsy: Subjects who received standard forceps biopsy either first or second during their biopsy of lung lesions.
  Standard forceps biopsy first, then crossover to receive the research cryoprobe biopsy during the procedure.
  Cryoprobe biopsy: A 1.1mm disposable cryoprobe that is passed through the working channel of the Ion Robotic bronchoscope to collect biopsy tissue
  Standard forceps biopsy: Biopsy forceps used to collect tissue
- Research Cryoprobe Biopsy First, Then Standard Forceps Biopsy: Subjects who received the research cryoprobe biopsy first or second during their biopsy of lung lesions.
  Research cryoprobe biopsy first, then crossover to receive the standard forceps biopsy during the procedure.
  Cryoprobe biopsy: A 1.1mm disposable cryoprobe that is passed through the working channel of the Ion Robotic bronchoscope to collect biopsy tissue
  Standard forceps biopsy: Biopsy forceps used to collect tissue
Period: First Intervention
Arm/Group | Standard Forceps Biopsy First, Then Research Cryoprobe Biopsy | Research Cryoprobe Biopsy First, Then Standard Forceps Biopsy
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Standard Forceps Biopsy First, Then Research Cryoprobe Biopsy | Research Cryoprobe Biopsy First, Then Standard Forceps Biopsy
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Forceps Biopsy First, Then Research Cryoprobe Biopsy | Research Cryoprobe Biopsy First, Then Standard Forceps Biopsy | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.3 (9.23) | 70.2 (7.11) | 70.3 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 7 | 11 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 15 | 13 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 15 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Ability to Successfully Obtain Sample
Description: Number of tissue samples that are considered by the bronchoscopist as adequate for further pathological analysis
Time Frame: Baseline
Measure: Number; unit: tissue samples
Groups:
- Standard Forceps Biopsy: Subjects who received standard forceps biopsy either first or second during their biopsy of lung lesions.
  Standard forceps biopsy: Biopsy forceps used to collect tissue
- Research Cryoprobe Biopsy: Subjects who received the research cryoprobe biopsy first or second during their biopsy of lung lesions.
  Cryoprobe biopsy: A 1.1mm disposable cryoprobe that is passed through the working channel of the Ion Robotic bronchoscope to collect biopsy tissue
Arm/Group | Standard Forceps Biopsy | Research Cryoprobe Biopsy
Number analyzed (Participants) | 30 | 30
tissue samples | 123 | 130

2. Secondary Outcome: Duration of Biopsy Procedure
Description: Total time of biopsy procedure from first insertion of probe into robotic sheath to removal of specimens.
Time Frame: Biopsy procedure, approximately 3 hours
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Standard Forceps Biopsy | Research Cryoprobe Biopsy
Number analyzed (Participants) | 30 | 30
minutes | 41 [30 to 53] | 41 [21 to 54]

3. Secondary Outcome: Freezing Time for Cryoprobe Biopsies
Description: Total freezing time for cryoprobe biopsies, measured in seconds
Time Frame: Biopsy procedure, approximately 60 seconds
Population: This outcome measure was only collected and analyzed for the Research cryoprobe biopsy arm
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Standard Forceps Biopsy | Research Cryoprobe Biopsy
Number analyzed (Participants) | 0 | 30
seconds |  | 4.54 (0.91)

4. Secondary Outcome: Number of Successful Biopsy Attempts
Description: One attempt is defined as insertion of the biopsy probe into the robotic sheath, activation/employment of the biopsy mechanism at the target site and retrieval via the robotic sheath. A biopsy attempt is successful if a tissue sample that is considered by the bronchoscopist to be adequate for further pathological analysis can be retrieved.
Time Frame: Biopsy procedure, approximately 3 hours
Measure: Number; unit: successful attempts
Arm/Group | Standard Forceps Biopsy | Research Cryoprobe Biopsy
Number analyzed (Participants) | 30 | 30
successful attempts | 123 | 130

5. Secondary Outcome: Histological Accessibility Grade
Description: Pathologic description ranging from insufficient to diagnostic material
Time Frame: Pathology review, approximately 1 day
Population: Data was not collected nor analyzed due to inadequate tissue size, volume, and quality, no data were collected for this Outcome Measure
Arm/Group | Standard Forceps Biopsy | Research Cryoprobe Biopsy
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Histological Diagnostic Yield
Description: Defined as the ability of the pathologist to make a diagnostic statement based on the histological analysis of the obtained tissue samples. Graded 1-4 with 1 being insufficient tissue and 4 being diagnostic material.
Time Frame: Pathology review, approximately 1 day
Population: as for outcome 5
Arm/Group | Standard Forceps Biopsy | Research Cryoprobe Biopsy
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Total Histological Area
Description: The total histological area of the biopsy samples. Measured in (mm^2)
Time Frame: Pathology review, approximately 1 day
Population: as for outcome 5
Arm/Group | Standard Forceps Biopsy | Research Cryoprobe Biopsy
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Crush Artifacts
Description: The total percent area of crush artifacts identified in the biopsy samples (percent total area)
Time Frame: Pathology review, approximately 1 day
Population: as for outcome 5
Arm/Group | Standard Forceps Biopsy | Research Cryoprobe Biopsy
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Other Pathologic Artifacts
Description: The total percent area of other pathologic artifacts identified in the tissue biopsy samples that obscure pathological assessment (percent total area)
Time Frame: Pathology review, approximately 1 day
Population: as for outcome 5
Arm/Group | Standard Forceps Biopsy | Research Cryoprobe Biopsy
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Different Tissue Types in the Tissue Specimen
Description: The total percent area of different tissue types identified in the tissue biopsy samples. Defined as the total of alveoli, bronchus, mucus, blood, and target tissue (percent total area)
Time Frame: Pathology review, approximately 1 day
Population: as for outcome 5
Arm/Group | Standard Forceps Biopsy | Research Cryoprobe Biopsy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each subject from baseline until completion of the standard of care post procedure follow-up for approximately 2 weeks
Arm/Group | Standard Forceps Biopsy | Research Cryoprobe Biopsy
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 3/30 | 2/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Forceps Biopsy (N=30) | Research Cryoprobe Biopsy (N=30)
Minor bleeding (Injury, poisoning and procedural complications) | 3 (3) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-15): https://cdn.clinicaltrials.gov/large-docs/82/NCT05399082/Prot_SAP_000.pdf